CLINICAL TRIAL: NCT03535922
Title: Evaluation of Routinely Measured PATtient Reported Outcomes in HemodialYsis Care (EMPATHY) Trial: A Cluster Randomized Controlled Trial
Brief Title: Evaluation of Routinely Measured Patient-reported Outcomes in Hemodialysis Care
Acronym: EMPATHY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RES0034066
Record Dates: First submitted 2018-04-30; First posted 2018-05-24 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Hemodialysis; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The disease-specific PROM group (Experimental): Hemodialysis (HD) units randomized to this PROMs assessment group will administer a disease-specific PROM every 2 months to all patients able to complete the instrument independently or with assistance for a period of 12 months. Patients will receive a copy of their PROM results in report form and patients will be prompted to follow-up with their care providers if they provide a positive response to any of the symptoms assessed by the PROM. The disease-specific PROM report will also be added to the patient's medical chart for review by clinicians. The report will display each patient's most recent results in comparison with their previous results, and in comparison with the general dialysis population. The PROM report will be accompanied by treatment aids for all symptoms. The proposed disease-specific PROM is the ESAS-r:Renal or the IPOS-Renal.
  Interventions: Other: PROMs Assessment
- The generic PROM group (Experimental): HD units randomized to this PROMs assessment group will administer a generic PROM every 2 months to all patients able to complete the instrument independently or with assistance for a period of 12 months. Patients will receive a copy of their PROM results in report form and patients will be prompted to follow-up with their care providers if they provide a positive response to any of the symptoms assessed by the PROM. The generic PROM report will also be added to the patient's medical chart for review by clinicians. The report will display each patient's most recent results in comparison with their previous results, and in comparison with the general dialysis population. The PROM report will be accompanied by treatment aids for all symptoms. The proposed generic PROM is the EQ-5D-5L.
  Interventions: Other: PROMs Assessment
- Disease-specific and generic PROMs group (Experimental): HD units randomized to this PROMs assessment group will administer a disease-specific and generic PROM every 2 months to all patients able to complete the instrument for a period of 12 months. Patients will receive a copy of both their PROMs results in report form and patients will be prompted to follow-up with their care providers if they provide a positive response to any of the symptoms assessed by the two PROMs. The disease-specific and generic PROMs reports will also be added to the patient's medical chart for review by clinicians. The report will display each patient's most recent results in comparison with their previous results, and in comparison with the general dialysis population. The PROMs reports will be accompanied by treatment aids for all symptoms.
  Interventions: Other: PROMs Assessment
- The control or 'usual care' group (No Intervention): HD units randomized to this group will follow usual care and patients will not have any PROMs assessment; however, all the treatment aids will be made available for clinicians in this study group during the 12 months trial period.

INTERVENTIONS:
Other: PROMs Assessment — Routine measurement and reporting of disease-specific PROMs, generic PROMs, or combination of both
  Arms: Disease-specific and generic PROMs group; The disease-specific PROM group; The generic PROM group

SUMMARY:
Patient-reported outcome measures (PROMs) are reports coming directly from patients about how they function or feel in relation to a health condition and its therapy, without interpretation of the patient's responses by a clinician or anyone else. PROMs capture patients' experiences of symptoms and impact of disease on functioning and can support clinicians to monitor disease progression and facilitate patient-centered care.

The EMPATHY trial will determine the effects of routinely measuring PROMs on the experiences of patients undergoing hemodialysis in Alberta and Ontario. In this study, two kinds of PROMs will be used: a disease-specific PROM and a generic PROM. The disease-specific PROM focuses on health symptoms related to kidney failure and the generic PROM focuses on general health.

In the trial, patients will be invited to complete the PROMs, and results of the measures will be linked to treatment aids for clinicians, providing specific information on how symptoms can best be managed. These care pathways will also be available to patients not receiving PROMs. The main outcome of this study will be patient-clinician communication, which will be assessed using a questionnaire called the "Communication Assessment Tool". In addition to assessing the effect of using these questionnaires on patient-provider communication, this study will allow us to explore whether their use affects patient management and symptoms, use of healthcare services, and the overall cost of implementing these questionnaires in clinical practice.

Each dialysis unit (including all patients) will be randomized to one of four study groups: 1) Patients will complete the disease-specific PROM; 2) Patients will complete the generic PROM; 3) Patients will complete both the disease-specific and generic PROM; 4) Patients will receive usual care.

Clinicians (in dialysis units randomized to PROMs, groups 1-3) will receive the results of the questionnaires completed by the patients. This is intended to trigger the clinician to ask the patient about certain symptoms if any exist. All clinicians in all study groups will have access to the clinical "treatment aids", which are tools that help identify and manage certain symptoms that patients might have. For example, people with severe itching will be cared for based on a step-wise treatment algorithm. Patients will also receive a report of their questionnaire(s) results, with an explanation of what it means.

DETAILED DESCRIPTION:
The overall aim of this study is to explore the usefulness of integrating PROM assessments in the clinical management of hemodialysis patients. The specific objectives are as follows:

Primary objective: to determine the effects of routine measurement and reporting to clinicians of PROMs, namely, the Edmonton Symptom Assessment System- revised: Renal (ESAS-r: Renal) or the Integrated Palliative care Outcome Scale - Renal (IPOS-Renal) and/or the EQ-5D-5L on patient-reported experience, particularly patient-clinician communication, measured by the Communication Assessment Tool (CAT), for patients with kidney failure requiring hemodialysis.

Secondary objectives:

1. To determine if there is a difference in patient-reported experience and other outcomes induced by a condition-specific (ESAS-r: Renal /IPOS-Renal) versus a generic (EQ-5D-5L) PROM;
2. To determine the effects of routinely measuring and reporting the ESAS-r: Renal/IPOS-Renal and/or the EQ-5D-5L on the clinical management of symptoms;
3. To determine the effects of routinely measuring and reporting the ESAS-r: Renal /IPOS-Renal and/or the EQ-5D-5L on overall HRQL;
4. To determine the effects of routinely measuring and reporting the ESAS-r: Renal/IPOS-Renal and/or the EQ-5D-5L on symptom burden, mental health outcomes and healthcare utilization;
5. To determine the cost-effectiveness of routinely measuring the ESAS-r: Renal/IPOS-Renal and/or the EQ-5D-5L for patients with kidney failure requiring hemodialysis;
6. To explore the perspectives and experience of patients and clinicians with routine measurement and reporting of PROMs in clinical practice.

Study Design:

The investigators propose the use of a cluster RCT design to avoid any potential contamination between the study groups. This study is a pragmatic RCT that will involve the random allocation of clusters (i.e., dialysis units) into four groups:

* Group 1: Completes disease-specific PROM
* Group 2: Completes generic PROM
* Group 3: Completes both PROMs
* Group 4: Usual care; does not complete any of the PROMs (control)

Treatment aids for symptoms assessed by the PROMs will be made available for all clinicians in all study groups. Details about intervention and treatment aids are provided below.

Hypotheses:

The investigators hypothesize that the routine measurement and reporting of PROMs will lead to improvement in communication between CKD patients and clinicians in dialysis units in Canada compared to usual care. The investigators also hypothesized that this will lead to better symptom and disease management, and improvement in mental health and quality of life. Furthermore, the investigators anticipate that this intervention will be cost-effective and will be acceptable and feasible in the dialysis units' environment.

Setting and Population:

All available dialysis units from Alberta (Alberta Kidney Care - North (AKC-N) and Alberta Kidney Care - South (AKC-S)) and selected units in Ontario (Ontario Renal Network - ORN) will be invited to participate in this study. The unit of randomization will be the dialysis units within AKC-N/AKC-S/ORN, not dialysis programs or individual patients. Randomization will be done within each renal program (AKC-N/AKC-S/ORN) to ensure that units from all programs are represented in all study groups.

Dialysis Unit Eligibility Criteria:

Inclusion Criteria:

* The unit provides chronic in-center hemodialysis;
* Hemodialysis clinicians are willing to review individual patients' routinely collected ESAS-r: Renal or IPOS-Renal and/or EQ-5D-5L as part of routine patient assessment;

Exclusion Criteria:

* The unit is unable to administer the ESAS-r: Renal or IPOS-Renal and EQ-5D-5L to in-centre hemodialysis patients as part of clinical workflow to all possible patients;
* The unit is part of a long-term care facility
* There are 5 or fewer patients treated at that unit
* Lack of WiFi connectivity (Alberta only)

Inclusion/exclusion criteria for individual patients: All patients undergoing hemodialysis who are 18 years or older at the start of the study, and are willing and able to complete the PROMs as part of the trial will be eligible to participate in this study. Patients with cognitive impairment, undergoing acute dialysis, or transiently dialyzing in the unit are not included.

Interventions:

Since blinding is not feasible in this trial, it will be conducted as an open trial. Consequently, research staff, clinicians, and all patients will be aware of group allocation; cluster randomization is intended to minimize potential biases associated with an open trial design. Eligible dialysis units will be randomly allocated to one of 4 study groups:

1. The disease-specific PROM group: The disease-specific PROM will be administered every 2 months to all patients able to complete the instrument for a period of 12 months. The PROMs results will be reported back to the patient, and patients will be prompted to follow-up with their care providers if they provide a positive response to any of the symptoms assessed by the PROM. The PROMs results will also be printed in a report form and added to the patient's medical chart for review by clinicians. The report will display each patient's most recent results in comparison with their previous results, and in comparison with the general dialysis population. The PROMs report will be accompanied by treatment aids for all symptoms.
2. The generic PROM group: The generic PROM will be administered every 2 months to all patients able to complete the instrument for a period of 12 months. The PROMs results will be reported back to the patient, and patients will be prompted to follow-up with their care providers if they provide a positive response to any of the symptoms assessed by the PROM. The PROMs results will also be printed in a report form and added to the patient's medical chart for review by clinicians. The report will display each patient's most recent results in comparison with their previous results, and in comparison with the general dialysis population. The PROMs report will be accompanied by treatment aids for all symptoms. The proposed generic PROM is the EQ-5D-5L.
3. The disease-specific and generic PROM group: The disease-specific and generic PROMs will be administered every 2 months to all patients able to complete the instrument for a period of 12 months. The PROMs results will be reported back to the patient, and patients will be prompted to follow-up with their care providers if they provide a positive response to any of the symptoms assessed by the PROM. The PROMs results will also be printed in a report form and added to the patient's medical chart for review by clinicians. The report will display each patient's most recent results in comparison with their previous results, and in comparison with the general dialysis population. The PROMs report will be accompanied by treatment aids for all symptoms.
4. The control or 'usual care' group: Patients in this group will follow usual care as provided in the dialysis unit and will not complete any PROM; however, all the treatment aids will be made available for clinicians in this study group during the trial period.

Treatment aids:

Treatment aids are assessment and treatment resources developed by expert clinicians for the management of certain symptoms and disorders. Each renal program developed treatment aids specific to symptoms assessed by the ESAS-r: Renal or IPOS-Renal (e.g., itchiness, restless leg syndrome, nausea) and the EQ-5D-5L (e.g., pain, anxiety/depression). Treatment aids are intended to support clinicians in the assessment and management of symptoms identified by these PROMs and will be made available for all clinicians at all study sites regardless of to which group they are randomized.

Patient-facing materials are also provided to patients, to help them better understand the reasons why their symptom/problem may have developed, treatment options that might be considered, as well as self-care activities they can undertake to alleviate the symptom or problem.

Data Analysis:

The primary analysis will assess change in the overall CAT score, between study groups from baseline to 12 months using a linear mixed-effects model, with the mean CAT for the dialysis unit at baseline as a fixed effect covariate, and dialysis unit (cluster) as a random intercept. Our primary analytic plan will be based on changes in mean CAT score at the unit level, from baseline to 12 months. The primary analysis will be based on all of the PROMs intervention groups combined compared to the control group as fixed effects. As one of our secondary objectives, assessing differences between specific and generic PROMs, we will compare the individual interventions groups (i.e., ESAS-r: Renal /IPOS alone, EQ-5D-5D alone, or the combination) to the control group.

We will also compare the proportion of patients reporting symptoms/problems on the ESAS-r: Renal or IPOS-Renal and EQ-5D-5L and the management of such symptoms/problems. Through clinical records, we will link PROMs scores with the use of specific treatments as per the treatment aids. We will obtain medication lists, allied health referrals, and chart notes to capture how symptoms are being treated. Each renal program (i.e., AKC-N, AKC-S, and ORN) will be analyzed separately then we will use meta-analyses to analyze the data from each renal program.

Economic Evaluation:

A cost-effectiveness analysis will be employed of the different study groups, compared to the usual care group as the reference case. The incremental costs and incremental QALYs of the different interventions relative to the usual care group will be compared to calculate incremental cost per QALYs gained ratios. Costs will be estimated for patients in the different study groups, including treatments received by patients, taking the perspective of the provincial health care system, personnel costs for training and delivery of the PROMs assessments, and subsequent health care utilization for patients in each of the study groups. Health care utilization will be estimated through linkage with provincial administrative health care databases at the individual patient-level. Costs associated with the provision of the intervention, including training and nursing time, will be estimated through observations for time and valued using standard staffing wage scales for the respective geographic regions. QALYs will be calculated based on changes in the EQ-5D-5L index score, using the Canadian preference weighting.

Study Period:

The study will be implemented over 48 months. The first 6 months will involve the administrative approvals, completing ethics requirements, training of clinicians on the use of PROMs; the following 18 months will involve trial implementation including assessments and interventions. The last 12-24 months will involve compiling the data from all study sites, data analysis and reporting of results.

ELIGIBILITY:
Inclusion criteria:

* Undergoing hemodialysis within an eligible in-centre dialysis unit in Alberta or Ontario
* 18 years or older at the start of the study
* Willing and able to complete the PROMs as part of the trial

Exclusion criteria:

* Cognitive impairment present
* Undergoing acute dialysis or transiently dialyzing in the unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3977 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Communication Assessment Tool (CAT) scores over 12 months | Measured at baseline, 6 months, and 12 months
  The CAT assesses patient perceptions of clinicians' interpersonal and communication skills. 'Communication' refers to the interactions between members of the healthcare team (i.e., nurses, nephrologists) and the patient.

SECONDARY OUTCOMES:
Change in EQ-5D-5L scores over 12 months | Measured at baseline, 6 months, and 12 months
  The EQ-5D-5L is a standardized generic measurement of health-related quality of life. This measure provides a simple descriptive profile and single index value for health status. The intended purpose of this measure for this survey is for clinical and economic evaluation of healthcare.
Change in Disease-specific PROM (ESAS or IPOS) scores over 12 months | Measured at baseline, 6 months, and 12 months
  Measure of symptom burden (choice of instrument depends on regional dialysis program). The purpose of this outcome measure is to enable tracking of the effectiveness of targeted symptom management strategies at the patient and program levels.
Symptom treatments initiated | 12 month study period
  Chart review for action taken as result of PROMs measurement
Change in GAD-2 scores over 12 months | Measured at baseline, 6 months, and 12 months
  Measured by the Generalized Anxiety Disorder 2 item questionnaire (GAD-2). The GAD-2 is a screening tool for anxiety.
Change in PHQ-2 scores over 12 months | Measured at baseline, 6 months, and 12 months
  Measured by the Patient Health Questionnaire- 2 items (PHQ-2). The PHQ-2 is a screening tool for depression.
Change in PACIC-11 scores over 12 months | Measured at baseline, 6 months, and 12 months
  The 'Patient Assessment of Chronic Illness Care-11 item questionnaire' measures a number of aspects of care, including patient activation; delivery system design and decision support; goal setting and tailoring; problem-solving and contextual counselling; follow-up and coordination.
Healthcare utilization over 12 months | One year prior and one year after the study intervention
  Survey and clinical data will be linked to administrative data on healthcare utilization of participants
Cost-effectiveness/cost-utility analysis | 12 month study period
  A cost-effectiveness analysis of the different study groups, compared to the usual care arm

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Johnson, PhD, Principal Investigator — University of Alberta
Locations (3):
- Canada (3):
  - Alberta Kidney Care - South, Calgary, Alberta
  - Alberta Kidney Care - North, Edmonton, Alberta
  - Ontario Renal Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boyce MB, Browne JP. Does providing feedback on patient-reported outcomes to healthcare professionals result in better outcomes for patients? A systematic review. Qual Life Res. 2013 Nov;22(9):2265-78. doi: 10.1007/s11136-013-0390-0. Epub 2013 Mar 17. PMID 23504544
- [Background] Marshall S, Haywood K, Fitzpatrick R. Impact of patient-reported outcome measures on routine practice: a structured review. J Eval Clin Pract. 2006 Oct;12(5):559-68. doi: 10.1111/j.1365-2753.2006.00650.x. PMID 16987118
- [Background] Valderas JM, Kotzeva A, Espallargues M, Guyatt G, Ferrans CE, Halyard MY, Revicki DA, Symonds T, Parada A, Alonso J. The impact of measuring patient-reported outcomes in clinical practice: a systematic review of the literature. Qual Life Res. 2008 Mar;17(2):179-93. doi: 10.1007/s11136-007-9295-0. Epub 2008 Jan 4. PMID 18175207
- [Background] Boyce MB, Browne JP, Greenhalgh J. The experiences of professionals with using information from patient-reported outcome measures to improve the quality of healthcare: a systematic review of qualitative research. BMJ Qual Saf. 2014 Jun;23(6):508-18. doi: 10.1136/bmjqs-2013-002524. Epub 2014 Feb 6. PMID 24505110
- [Background] Antunes B, Harding R, Higginson IJ; EUROIMPACT. Implementing patient-reported outcome measures in palliative care clinical practice: a systematic review of facilitators and barriers. Palliat Med. 2014 Feb;28(2):158-75. doi: 10.1177/0269216313491619. Epub 2013 Jun 25. PMID 23801463
- [Background] Patrick DL, Deyo RA. Generic and disease-specific measures in assessing health status and quality of life. Med Care. 1989 Mar;27(3 Suppl):S217-32. doi: 10.1097/00005650-198903001-00018. PMID 2646490
- [Background] Laupacis A, Wong C, Churchill D. The use of generic and specific quality-of-life measures in hemodialysis patients treated with erythropoietin. The Canadian Erythropoietin Study Group. Control Clin Trials. 1991 Aug;12(4 Suppl):168S-179S. doi: 10.1016/s0197-2456(05)80021-2. PMID 1663853
- [Background] Perrone RD, Coons SJ, Cavanaugh K, Finkelstein F, Meyer KB. Patient-reported outcomes in clinical trials of CKD-related therapies: report of a symposium sponsored by the national kidney foundation and the U.S. Food and Drug Administration. Am J Kidney Dis. 2013 Dec;62(6):1046-57. doi: 10.1053/j.ajkd.2013.07.004. Epub 2013 Aug 26. PMID 23988757
- [Background] Davison SN, Jhangri GS, Johnson JA. Longitudinal validation of a modified Edmonton symptom assessment system (ESAS) in haemodialysis patients. Nephrol Dial Transplant. 2006 Nov;21(11):3189-95. doi: 10.1093/ndt/gfl380. Epub 2006 Sep 6. PMID 16957010
- [Background] Fayers PM. Evaluating the effectiveness of using PROs in clinical practice: a role for cluster-randomised trials. Qual Life Res. 2008 Dec;17(10):1315-21. doi: 10.1007/s11136-008-9391-9. Epub 2008 Sep 27. PMID 18821031
- [Derived] Johnson JA, Al Sayah F, Buzinski R, Corradetti B, Davison SN, Elliott MJ, Klarenbach S, Manns B, Schick-Makaroff K, Short H, Thomas C, Walsh M. A cluster randomized controlled trial for the Evaluation of routinely Measured PATient reported outcomes in HemodialYsis care (EMPATHY): a study protocol. BMC Health Serv Res. 2020 Aug 10;20(1):731. doi: 10.1186/s12913-020-05557-z. PMID 32778102